CLINICAL TRIAL: NCT04575129
Title: Cross-cultural Adaptation, Reliability, and Validity of Self Administered Neck Mobility Assessment Tool (S-ROM-Neck): Turkish Version
Brief Title: Psychometric Properties of the Turkish Version of S-ROM-Neck
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Emine Aslan Telci, Principal Investigator, Pamukkale University
Other Study IDs: S-ROM-Neck
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Neck Pain
Keywords: Surveys and Questionnaires; Neck Pain; Range of Motion; Psychometrics
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: No intervention will be applied
  Interventions: Other: No intervention will be applied

INTERVENTIONS:
Other: No intervention will be applied — No intervention will be applied

SUMMARY:
Patient-reported joint motion assessment tools have been developed and applied successfully in several joints of the body. "The Self Administered Neck Mobility Assessment Tool (S-ROM-Neck)" questionnaire was developed by Langenfeld et al in 2018. With this questionnaire, the clinicians are able to evaluate the neck joint motion perception of the patients, subjectively. There is no Turkish version of the questionnaire. The aim of our study is to develop the Turkish version of the S-ROM-Neck questionnaire, to analyze its cultural adaptation, and to reveal its validity and reliability.

DETAILED DESCRIPTION:
Neck pain leads to a decreased range of motion in the cervical spine, bringing along functional losses. As a result, this situation is associated with many disabilities. Evaluation of neck joint motion is essential in patients with chronic neck pain. It is used to evaluate the neck pain level and functional deficit level of the patient. In this way, it is possible to evaluate the effectiveness of the treatment applied to the patient during the rehabilitation process. Generally, this evaluation can be made and interpreted by an experienced clinician. However, patient perception provides a better understanding of patients' needs and problems by converting clinical data into a patient-centered measure. Moreover, the patient's perspective can add valuable information to the examination by creating a holistic picture of the patient's problems, possible needs, and expectations. In 2018, the "Self Administered Neck Mobility Assessment Tool (S-ROM-Neck)" survey was developed by Langenfeld et al. With this questionnaire, developers purposed to evaluate the neck joint motion perception of the patients, subjectively. There is no Turkish version of the questionnaire. The aim of our study is to develop the Turkish version of the S-ROM-Neck questionnaire, to analyze its cultural adaptation, and to reveal its validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* To have neck pain for at least 3 months.
* Turkish literate individual

Exclusion Criteria:

* Operation history due to neck pain problems
* Individuals diagnosed with tumor, infection, ankylosing spondylitis, rheumatoid arthritis or inflammatory diseases, fracture, cauda equina syndrome
* Pregnancy
* Individuals who do not give consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
S-ROM-Neck | 5 minutes
  The scale includes six questions that target the primary movements of the neck joint (i.e. flexion, extension, rotation, and lateral flexion). Patients are asked to actively perform each neck movement and then rate the restriction they perceive during movement. This is done for each of the 6 directions of motion. Perceived restriction may be due to pain, stiffness, and/or tension. S-ROM-Neck has a structure scored with a visual analog scale (VAS). The left side contains the words "none" to indicate severe ROM restriction and the right side "as far as I want" to indicate maximum ROM. Explanatory pictures accompany each question. The total score is calculated by adding individual scores (minimum score [600] = no restriction; maximum score [0] = total restriction).

SECONDARY OUTCOMES:
Visual Analog Scale | 2 minutes
  It is scored between 0 and 10. While 0 indicates no pain, 10 indicates the most severe pain. With this scale, which is frequently used in individuals with chronic low back pain, the resting and activity pain of the individuals will be questioned.
Neck Disability Index | 5 minutes
  The Neck Disability Index consists of 10 sections: pain intensity, personal care, weight lifting, reading, headaches, concentration, work-life, driving, sleep and leisure activities. Each segment has a value ranging from zero (positive case) to five points (negative state). The total score on the Neck Disability Index ranges from zero to 50, and the high score corresponds to high disability.
Neck range of motion (ROM) measurement with inclinometer | 10 minutes
  Cervical region flexion, extension, lateral flexion and rotation movements will be evaluated with a Baseline Bubble Inclinometer. The inclinometer is a valid and reliable method for evaluating the cervical range of motion (14). While evaluating the flexion, extension and lateral flexion movements in the cervical region with the inclinometer, it was placed at the top of the head as the pivot point and the participant will be asked to perform the movement to the endpoint and return to the previous position. For rotation movement, the inclinometer will be placed on the participant's forehead in the supine position, and rotation movement will be requested from the patient. The value measured in the inclinometer will be recorded. Each move will be evaluated 3 times separately and its average will be noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University Hospital, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided